CLINICAL TRIAL: NCT02763865
Title: A Pilot Study to Assess the Effects of Pre-SMA LF-rTMS for the Treatment of Essential
Brief Title: A Pilot Study to Assess the Effects of Pre-SMA LF-rTMS for the Treatment of Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00033680
Record Dates: First submitted 2016-04-12; First posted 2016-05-05 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active pre-SMA rTMS (Experimental): The intervention to be administered is the MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil l to administer active rTMS at 1Hz, 1,200sec, 110% resting motor threshold (rMT); 1200 pulses total. Two Thymapad Stimulus Electrodes will be placed in the appropriate position during active rTMS administration.This intervention method will be used for all 15 treatment sessions (20 minutes/session).
  Interventions: Device: MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil
- Sham pre-SMA rTMS (Sham Comparator): The intervention to be administered is the eSHAM system used in conjunction with the MagVenture MagProx100 Stimulator with the Cool-B65 A/P Coil. For eSHAM administration two Thymapad Stimulus Electrodes will be placed on the scalp location that corresponded to left DLPFC. This intervention method will be used for all 15 treatment sessions (20 minutes/session). Previous studies have shown the eSHAM system effectively blinds participants to rTMS treatment (active versus sham).
  Interventions: Device: eSHAM system

INTERVENTIONS:
Device: MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil — Active rTMS administration (1Hz, 1,200sec, 110% resting motor threshold (rMT); 1200 pulses total.
  Resting motor threshold assessment the TMS machine will initially be set to 50% of its maximal output.
  Arms: Active pre-SMA rTMS
Device: eSHAM system — implemented in conjunction with the Cool-B65 A/P coil to effectively blind participants to rTMS treatment (active or sham)
  Arms: Sham pre-SMA rTMS

SUMMARY:
The purpose of this study is to determine the effects of Low Frequency Repetitive Transcranial Magnetic Stimulation (LF r-TMS) of the pre-Supplementary Motor Area (pre-SMA) on tremor as measured by the tremor rating scale (TRS) in patients with Essential Tremor (ET).

Hypothesis: Pre-SMA LF r-TMS will result in a >30% reduction in tremor as measured by the TRS. Another purpose of this study is to identify the mechanism by which LF r-TMS of the pre-SMA effects tremor in patients with ET.

Hypothesis: Inhibition of the pre-SMA by LF r-TMS improves tremor in ET by normalizing pre-SMA output, and improving motor control, as determined shortening of the delay in the second agonist burst, seen in ET patients. At conclusion of this study expect to have sufficient pilot data to justify larger pivotal trials designed to establish the efficacy of pre-SMA r-TMS in ET.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 of age
* Meet the diagnostic criteria for essential tremor with visible upper limb tremor
* Must be either on stable medications to treat tremor for 30 days, or no medications to treat tremor

Exclusion Criteria:

* History of seizures
* History of chronic pain conditions
* Any metal in their body above their shoulders
* Use of medications that lower seizure threshold including:

  * broad classes of drugs such as tricyclic antidepressants
  * anti-psychotics
  * neuroeptics
  * thyroid medications and stimulants
* Use of any medications that cause tremor, Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2017-03-21 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: clinic
Pre-assignment Details: screening procedures per inclusion and exclusion criteria, no wash out, stayed on meds.
Groups:
- Active: Active pre-SMA rTMS
- Sham: sham tms
Period: Overall Study
Arm/Group | Active | Sham
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: active tms
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (12.17) | 71.6 (12.17) | 71.6 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Mean TRS at Baseline Visit [Mean (Standard Deviation); unit: units on a scale] — TRS scale is a range of 0 - 84 (0 being the least severe and 84 being the most severe tremor)
  units on a scale | 36.0 (8.276) | 34 (5.385) | 35 (6.667)

OUTCOME MEASURES:

1. Primary Outcome: Mean TRS (Tremor Rating Score)
Description: Participants will be videotaped as they are being examined for the purpose of rating their tremor for the TRS. TRS scale is a range of 0 - 84 (0 being the least severe and 84 being the most severe tremor)
Time Frame: Baseline (Visit 2) post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 5
units on a scale | 26.6 (7.701) | 27.6 (8.325)

2. Primary Outcome: Mean TRS (Tremor Rating Score) at 4 Week Followup
Description: as for outcome 1
Time Frame: 4 week followup(visit 18)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 5
units on a scale | 29.60 (9.555) | 29.2 (5.891)

3. Primary Outcome: Mean TRS (Tremor Rating Score) at 8 Week Followup
Description: as for outcome 1
Time Frame: 8 week followup (visit 19)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham Pre-SMA rTMS: The intervention to be administered is the eSHAM system used in conjunction with the MagVenture MagProx100 Stimulator with the Cool-B65 A/P Coil. For eSHAM administration two Thymapad Stimulus Electrodes will be placed on the scalp location that corresponded to left DLPFC. This intervention method will be used for all 15 treatment sessions (20 minutes/session). Previous studies have shown the eSHAM system effectively blinds participants to rTMS treatment (active versus sham).
  MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil: Active rTMS administration (1Hz, 1,200sec, 110% resting motor threshold (rMT); 1200 pulses total.
  Resting motor threshold assessment the TMS machine will initially be set to 50% of its maximal output.
  eSHAM system: implemented in conjunction with the Cool-B65 A/P coil to effectively blind participants to rTMS treatment (active or sham)
Arm/Group | Active Pre-SMA rTMS | Sham Pre-SMA rTMS
Number analyzed (Participants) | 5 | 5
units on a scale | 29.6 (9.555) | 29.6 (5.771)

4. Primary Outcome: Mean TRS (Tremor Rating Score) at 12 Week Followup
Description: as for outcome 1
Time Frame: 12-week followup(visit 20)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 5
units on a scale | 32.8 (7.294) | 29.6 (8.264)

ADVERSE EVENTS:
Groups:
- Active Pre-SMA rTMS: The intervention to be administered is the MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil l to administer active rTMS at 1Hz, 1,200sec, 110% resting motor threshold (rMT); 1200 pulses total. Two Thymapad Stimulus Electrodes will be placed in the appropriate position during active rTMS administration.This intervention method will be used for all 15 treatment sessions (20 minutes/session).
  MagVenture MagProx100 Stimulator with a Cool-B65 A/P coil: Active rTMS administration (1Hz, 1,200sec, 110% resting motor threshold (rMT); 1200 pulses total.
  Resting motor threshold assessment the TMS machine will initially be set to 50% of its maximal output.
Arm/Group | Active Pre-SMA rTMS | Sham Pre-SMA rTMS
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes